CLINICAL TRIAL: NCT00136591
Title: A Phase 2 Study of Velcade™ in Subjects With Relapsed or Refractory Follicular B-Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: An arm closed due to lack of efficacy
Sponsor: Lymphoma Study Association (Other)
Collaborators: Janssen-Cilag International NV (Industry)
Responsible Party: B Coiffier, GELA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FL05-1; Janssen: 28866138-LYM-2003; Eudrac: 2005-000734-21
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma; bortezomib; relapse
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Arm A: a 21-day cycle of 1.5 mg/m2 Velcade™ twice weekly for 2 weeks. Days 1, 4, 8, and 11 of a 21-day cycle. Subjects in this treatment arm will receive a total of 8 cycles of treatment,
  Interventions: Drug: Bortezomib
- B (Experimental)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Arm A: a 21-day cycle of 1.5 mg/m2 Velcade™ twice weekly for 2 weeks. Days 1, 4, 8, and 11 of a 21-day cycle
  Arms: A
Drug: Bortezomib — Arm B: a 35-day cycle of 1.6 mg/m2 Velcade™once weekly for 4 weeks. Days 1, 8, 15, and 22 of a 35-day cycle. Subjects in this treatment arm will receive a total of 6 cycles of treatment, approximately 30 weeks.
  Arms: B

SUMMARY:
This is a prospective, randomized, sequential, international, multicentric, 2-arm, non-comparative, open-label, 2-stage clinical study to determine disease response rates to Velcade™ therapy in subjects who have relapsed or refractory follicular B-cell lymphoma.

Qualitative comparisons of the 2 treatment arms based on safety, efficacy and dosing convenience will be made in order to recommend a dose schedule for further clinical study.

DETAILED DESCRIPTION:
This is a prospective, randomized, sequential, international, multicentric, 2-arm, non-comparative, open-label, 2-stage clinical study to determine disease response rates therapy of Velcade™ in subjects who have relapsed or refractory follicular B-cell lymphoma (FLL).

Qualitative comparisons of the 2 treatment arms based on safety, efficacy and dosing convenience will be made in order to recommend a dose schedule for further clinical study.

It is anticipated that approximatively 120 subjects will be enrolled to achieve the required 110 evaluable subjects, 55 in each treatment arm. Patients who receive any amount of Velcade™ are evaluable. Subjects not evaluable for response will be replaced.

A central randomization will be used in this study. Subjects will be randomized and stratified with factors for prior therapies (1 or 2 versus > 2) and time to progression (TPP) for the last given anti-neoplastic therapy (≤ 12 months versus > 12 months).

The eligible subjects will be randomized to either Treatment Arm A or Treatment Arm B in a 1:1 ratio:

* Subjects randomized to Treatment Arm A will receive 1.5 mg/m² Velcade™ administered biweekly on Days 1, 4, 8, and 11 of a 21-day cycle. Patients will receive 8 cycles. The dose of Velcade™ received in schedule A will be 48 mg/m² over 24 weeks.
* Subjects randomized to Treatment Arm B will receive 1.6 mg/m² Velcade™ administered weekly on Days 1, 8, 15, and 22 of a 35-day cycle. Patients will receive 6 cycles. The dose of Velcade™ received in schedule B will be 38.4 mg/m² over 30 weeks.

Two additional cycles may be administered if the patient shows improvement to PR after 8 or 6 cycles for arm A or B, respectively.

Study drug dose and schedule reduction for toxicity will be allowed during the study.

A two stage interim analysis will be conducted in each treatment arm to determine whether either of the 2 treatments lacks sufficient efficacy.

The final analysis will be conducted when all subjects have had the opportunity to complete the 30 day post-treatment evaluation visit. All data from all visits up until this point will be used in the final analysis, including data from any follow-up visits that have occurred.

Patients will be recruited approximately over 2 years and followed until all data are available for final analysis.

The total duration of the study is expected to be 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 18 years or older.
* Initial diagnosis of follicular B-cell lymphoma (CD20+) (grades 1, 2, and 3 based on the World Health Organization 1997 classification), in first or subsequent relapse or progression after prior anti-neoplastic treatment including previous rituximab treatment. Relapse or progression since previous anti-neoplastic therapy must be documented by new lesions or objective evidence of progression of existing lesions.
* At least 1 measurable lymph node mass that is >1.5 cm in 2 perpendicular dimensions, and has not been previously irradiated or has grown since previous irradiation.
* No active central nervous system (CNS) lymphoma
* Karnofsky Performance Status (KPS) >50% (Eastern Cooperative Oncology Group [ECOG] 0-2)
* The following laboratory values at screening, unless abnormalities are related to the lymphoma:

  * Absolute neutrophil count (ANC) >1000 cells/dL;
  * Platelets >50,000 cells/dL;
  * Aspartate transaminase (AST) <3 x upper limit of normal (ULN);
  * Alanine transaminase (ALT) <3 x ULN;
  * Total bilirubin <2 x ULN;
  * Creatinine level <150 µmol/L
* Toxic effects of previous therapy or surgery resolved to Grade 2 or better.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Women are neither breast feeding nor pregnant for the duration of the study. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women. Male subject agrees to use an acceptable method of contraception for the duration of the study.
* Voluntary signed informed consent before performance of any study-related procedure not part of normal medical care.
* Patient with minimum life expectancy of 3 months.

Exclusion Criteria:

* Any other type of lymphoma.
* Previous treatment with Velcade™.
* Anti-neoplastic or experimental or radiation therapy within 3 weeks before Day 1 of Cycle 1.
* Major surgery within 2 weeks before Day 1 of Cycle 1.
* Rituximab, alemtuzumab (Mabcampath®), or other unconjugated therapeutic antibody within 10 weeks before Day 1 of Cycle 1.
* Nitrosoureas within 6 weeks before Day 1 of Cycle 1.
* Radioimmunoconjugates or toxin immunoconjugates such as ibritumomab tiuxetan (Zevalin™), or tositumomab (Bexxar®) within 10 weeks before Day 1 of Cycle 1.
* Peripheral neuropathy or neuropathic pain of Grade 3 or worse.
* History of allergic reaction attributable to compounds containing boron or mannitol.
* Diagnosed or treated for a malignancy other than non-Hodgkin's lymphoma (NHL) within 5 years before Day 1 of Cycle 1, with the exception of complete resection of basal cell carcinoma, squamous cell carcinoma of the skin, or in situ malignancy.
* Active systemic infection requiring treatment.
* Previously known HIV positive serology.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Concurrent treatment with another investigational agent.
* Adult patient under guardian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2005-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine the response rate to Velcade™ as a single agent | End of treatment

SECONDARY OUTCOMES:
To determine the overall complete response (CR) rate (CR + complete response unconfirmed [CRu]) | End of treatment
To determine time to progression (TTP) | End of study
To determine overall survival | End of study
To determine duration of response | End of study
To determine the time to best response | End of study
To evaluate the safety and tolerability of Velcade™ | End of study
To evaluate the effects of Velcade™ given biweekly at 1.5 mg/m2 versus 1.6 mg/m2 weekly | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Coiffier, MD, Study Chair — Hospices Civils de Lyon, Lyon, France; Vincent Ribrag, MD, Principal Investigator — Institut Gustave Roussy, Villejuif, France
Locations (4):
- Groupe d'Etude des Lymphomes de l'adulte, Mont-Godinne, Belgium
- France (3):
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] O'Connor OA, Wright J, Moskowitz C, Muzzy J, MacGregor-Cortelli B, Stubblefield M, Straus D, Portlock C, Hamlin P, Choi E, Dumetrescu O, Esseltine D, Trehu E, Adams J, Schenkein D, Zelenetz AD. Phase II clinical experience with the novel proteasome inhibitor bortezomib in patients with indolent non-Hodgkin's lymphoma and mantle cell lymphoma. J Clin Oncol. 2005 Feb 1;23(4):676-84. doi: 10.1200/JCO.2005.02.050. Epub 2004 Dec 21. PMID 15613699
- [Background] Goy A, Younes A, McLaughlin P, Pro B, Romaguera JE, Hagemeister F, Fayad L, Dang NH, Samaniego F, Wang M, Broglio K, Samuels B, Gilles F, Sarris AH, Hart S, Trehu E, Schenkein D, Cabanillas F, Rodriguez AM. Phase II study of proteasome inhibitor bortezomib in relapsed or refractory B-cell non-Hodgkin's lymphoma. J Clin Oncol. 2005 Feb 1;23(4):667-75. doi: 10.1200/JCO.2005.03.108. Epub 2004 Dec 21. PMID 15613697
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In french) — http://www.gela.org